CLINICAL TRIAL: NCT06014892
Title: The 4th Trimester Initiative: The Impact of Parental Support on Pregnant Trainee Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Brigham and Women's Hospital (Other); Boston Children's Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Erika Rangel, MD, Associate Surgeon, Assistant Professor of Surgery, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2022P001157
Record Dates: First submitted 2023-08-11; First posted 2023-08-28 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Pregnancy Related; Burnout, Professional; Wellness, Psychological
Keywords: burnout; postpartum depression; lactation; resident attrition
MeSH Terms: conditions — Burnout, Professional; Psychological Well-Being; Burnout, Psychological; Depression, Postpartum; Breast Feeding

STUDY DESIGN:
Intervention Model Description: This study is designed as a prospective randomized open-labeled study. We plan to enroll 152 trainees who are pregnant or immediately post-partum. Participants will undergo stratified randomization to an intervention or no intervention arm in a 1 to 1 ratio based on training specialty (either procedural or non-procedural) and training site (MGH, BWH, BCH, or BIDMC). Procedural specialties are defined as specialties that spend a significant portion of their training performing procedures: this includes all surgical specialties, anesthesiologists, gastroenterologists, obstetricians-gynecologists, interventional-radiologist, interventional-pulmonologists, interventional-cardiologists, emergency physicians. All other training programs are considered non-procedural specialties.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group will receive:
  1. A Snoo smart sleep bassinet
  2. A Willow wearable breast pump
  3. Access to Maven Clinic for 24/7 on-demand perinatal care
  4. A faculty mentor in their own department
  Interventions: Device: Snoo smart bassinet; Device: Willow wearable breast pump; Behavioral: Maven Clinic on-demand perinatal consultation; Behavioral: Faculty mentor
- Control (No Intervention): The control arm will receive:
  Current standard in the residency training program.

INTERVENTIONS:
Device: Snoo smart bassinet — Participants in the intervention arm will be shipped a Snoo bassinet during their third trimester. The bassinet must be returned to the company at 6 months
  Arms: Intervention
Device: Willow wearable breast pump — Participants in the intervention arm will be shipped a Willow wearable breast pump and milk storage bags during the third trimester, which participants may keep
  Arms: Intervention
Behavioral: Maven Clinic on-demand perinatal consultation — Participants in the intervention arm will receive immediate access to Maven Clinic for 24/7 on-demand consultation with perinatal specialists.
  Arms: Intervention
Behavioral: Faculty mentor — After enrollment, participants in the intervention arm will be paired with a faculty mentor who is also a mother to discuss issues related to work-family integration during pregnancy and early infancy.
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to determine the impact of a parental support package for new trainee mothers which focuses on mentorship, lactation, and sleep, and access to perinatal care. The main questions it aims to answer are whether this set of interventions will improve trainee wellbeing and decrease medical error.

Participants will be randomized to intervention and control groups. The intervention group will receive:

1. A Snoo smart sleep bassinet
2. A Willow wearable breast pump
3. Access to Maven Clinic for 24/7 on-demand perinatal care
4. A faculty mentor in their own department

The control group will receive the standard support currently offered by training programs.

All participants will wear a Fitbit to track sleep and will take a series of surveys querying pregnancy, birth, and postpartum experiences; wellbeing; and professional satisfaction.

Researchers will compare intervention and control groups to see if the intervention group has:

1. decreased rates of burnout
2. increased professional fulfillment
3. decreased thoughts of leaving the profession
4. increased perception of organizational and personal value alignment
5. increased sleep
6. decreased risk of medical errors
7. increased personal fulfillment of breastfeeding goals
8. decreased risk of postpartum depression

DETAILED DESCRIPTION:
The birth of a child during training is a significant life event that has been associated with a high risk of attrition and career dissatisfaction. Post-graduate training lasts between 3 and 9 years after medical school and overlaps with peak child-bearing years. The difficulties facing new trainee parents have been characterized with stigma, health concerns due to unmitigated work schedules during pregnancy, short parental leaves, and challenges with lactation and childcare contributing to stress and fatigue. Program directors describe marked variability in how childbearing affected residents' quality of work, with many describing returning residents as conflicted and distracted. The increase in family commitments in the setting of existing training demands can lead trainees to develop a perception of work-life incompatibility, fatigue, to change their career trajectory, and to have increased risk of burnout and postpartum depression. The investigators hypothesize that a set of interventions for new trainee mothers, focusing on mentorship, lactation, and sleep can improve trainee wellbeing and decrease the risk of medical errors.

STUDY PROCEDURES:

This study is designed as a prospective randomized clinical trial of pregnant trainees at Massachusetts General Hospital (MGH), Brigham and Women's Hospital (BWH), Boston Children's Hospital (BCH), and Beth Israel Deaconess Medical Center (BIDMC).

Participants will be screened over the phone and consent to participate obtained in person. All participants will take the electronic pre-intervention assessment survey after consent. After completion of the pre-intervention assessment survey, participants will be randomized into either the control arm or the intervention arm and provided a wearable device to monitor sleep (for one week during pregnancy to establish a baseline and for 6 months after delivery).

After delivery, all participants will take a set of surveys at 4,12,16,20,24, and 52 weeks postpartum querying obstetric and postpartum experiences; self-reported medical error; fatigue; wellbeing; and professional satisfaction.

The intervention group will receive:

1. A Snoo smart sleep bassinet
2. A Willow wearable breast pump
3. Access to Maven Clinic for 24/7 on-demand perinatal care
4. A faculty mentor in their own department

The control group will receive standard parental support currently offered by training programs.

Researchers will compare the following between intervention and control groups:

1. burnout
2. professional fulfillment
3. thoughts of leaving the profession
4. perception of organizational and personal value alignment
5. sleep and fatigue
6. self-reported medical errors
7. personal fulfillment of breastfeeding goals
8. risk of postpartum depression

The investigators plan to measure mean scores in burnout as our primary outcome. An effect size of 0.5 standard deviation change in burnout between the control and intervention arm is estimated to be a clinically relevant change. Trainees have mean burnout scores of 3.35 (SD=2.05). 76 subjects in each arm are estimated to be needed, 152 participants total, to detect a statistically significant change in burnout score (by at least 1.025 using the SPFI), with 80% power with a two tailed alpha of 10%, and allowing for 20% attrition of study subjects.

STATISTICAL ANALYSIS The investigators plan to report descriptive data including frequency, mean (SD) and median (inter-quartile range) for all outcome measures, using chi-squared analyses for categorical variables and t-test for continuous variables.

Mass General Brigham (MGB) has more than 200 training programs across its training sites. Of the 27/200+ programs that responded to a brief survey through the Wellbeing Council, 76 trainees (43 men and 33 women) became new parents this past academic year (2020-2021). Human Resources at MGB estimates more than 70 trainees apply for formal parental leave yearly which likely significantly underestimates the true number of new parents as most nonchildbearing parent trainees do not take formal parental leave. Based on this information, the investigators anticipate that the MGB training programs alone will have a sufficient number of trainees to conduct this study.

STUDY TERMINATION CRITERIA:

The study will be terminated at the request of the participant for any reason. Otherwise, the study will be terminated at 6 months. Subjects in the control arm who purchase a SNOO bassinet or a wearable breast pump will be requested to notify the study PI and will be categorized as a subgroup and analyzed in a planned sub-group analysis.

MONITORING AND QUALITY ASSURANCE:

To minimize the risk of loss of anonymity, participants will be assigned a unique study identifier. Access to files linking identifiers with identifying coded data will be limited only to need-to-know study personnel and stored in a Partners Password Protected online storage drive, while survey data will be obtained using Partners REDCap. Data will be accessible only to the PI and CITI-certified research staff. The Research staff will review the database each time new patient data is collected using a Partners password-protected computer and the PI will review the database once a month with details discussed at a monthly research meeting.

Identifying information (name, email address, phone number, shipping address, and due date) will need to be released to the sponsoring companies to facilitate delivery of the automated bassinet (Happiest Baby Inc), wearable breast pump (Willow Innovations) and access to perinatal on-demand consultation (Maven Clinic). Data transfer will be performed via MGB approved password protected and encrypted mechanisms. Both companies have designated representatives that are HIPAA certified with no association to the study execution or analysis. Data access by the company representatives will require multi-factor identification for the single user who will be allowed access. The transferred information will be used to order study related equipment for participants. The data will be deleted from the secure electronic location at the conclusion of the study.

Sleep tracking data is housed in secure Azure (Microsoft) servers. Fitabase uses Secure Sockets Layer (SSL) for all authentication (logins), billing, and administration of the site. The user's browser establishes the authenticity by requesting an SSL certificate that verifies the identity of Fitabase. Once that SSL certificate is recognized, a Secure Sockets Layer (SSL) connection is established for security, encrypting data transmitted between browser and web server.

Participants will be asked in person or online to authorize use of Fitabase to access their wearable device data and make it available for download for analysis. Participants will be informed that research staff will be able to access, view, and download deidentified data through the Fitabase platform. Data collected will relate to sleep length, movement, and quality. There are two instances when the PI will revoke access to data associated with participants in this study. First, if a participant chooses to withdraw from the study, the PI will remove the participant from the study platform (Fitabase) and data will be removed from the study. Second, 90 days after the completion of data collection Fitabase will remove the project from their data management system, disassociate the data from the project, and begin remove access to the data by deleting it from its servers and backup systems.

The PI will be responsible for determining whether the research should be altered or stopped. Throughout the duration of the study, the PI will perform ongoing evaluation of subject safety data to identify adverse events and trends as soon as possible. Any unanticipated adverse events involving risk to human subjects will be reviewed by the Principal Investigator and will be quickly reported to the Human Research Committee within the required time frame and to all participating investigators by The PI according to the Partners Human Research Committee guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Currently pregnant
* Part of a residency or fellowship training program at MGH, BWH, BCH, or BIDMC during pregnancy and for 6 months postpartum
* Clinically active and will remain clinically active until 6 months postpartum

Exclusion Criteria:

* significant cardiopulmonary, gastrointestinal, or neurologic comorbidities in participant or her fetus
* on research elective or dedicated research time from time of enrollment until 6 months postpartum.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2023-05-25 (Actual); Primary Completion 2026-01-25 (Actual); Study Completion 2026-01-25 (Actual)

PRIMARY OUTCOMES:
Burnout measured by emotional exhaustion and Interpersonal Disengagement components of the Stanford Professional Fulfillment Index | At Enrollment; 16 weeks postpartum; 24 weeks postpartum
  Emotional exhaustion and Interpersonal Disengagement are EACH scored on a scale of 0-10; The Emotional Exhaustion and Interpersonal Disengagement Scores are then averaged for score 0-10. Higher scores indicate higher likelihood of emotional exhaustion, interpersonal disengagement, and burnout (higher score is worse outcome)

SECONDARY OUTCOMES:
Professional Fulfillment measured by the Stanford Professional Fulfillment Index | At Enrollment; 16 weeks postpartum; 24 weeks postpartum; 1 year postpartum
  Professional Fulfillment is score on a scale of 0-10 with higher scores indicating a higher likelihood of professional fulfillment (higher score is better outcome)
Self reported medical error resulting in patient harm | 4 weeks, 12 weeks, 16 weeks, 20 weeks, and 24 weeks postpartum
  Participants will be asked "Over the past 4 weeks, how many times did you make a medical error that did result in patient harm?". Participants will be given options of "0", "1", "2", "3", or "3 or more".
Self reported medical error resulting in near miss for patient harm | 4 weeks, 12 weeks, 16 weeks, 20 weeks, and 24 weeks postpartum
  Participants will be asked "Over the past 4 weeks, how many times did you make a medical error that could have resulted in patient harm?". Participants will be given options of "0", "1", "2", "3", or "3 or more".
Organizational and Personal Values Alignment | At Enrollment; 16 weeks postpartum; 24 weeks postpartum
  3-item Stanford Values Alignment Scale. This validated instrument contains 3 statements with which participants are asked to indicate their agreement on a 5-point Likert Scale (0=not at all true; 4=completely true). Aggregate scores are determined by summing the 0-4 score of the individual items to yield a total score ranging from 0-12. Higher values are positive (indicate better alignment between organizational and personal values).
Negative Impact of Work on Personal Relationships | At Enrollment; 16 weeks postpartum; 24 weeks postpartum
  4-item Impact of Work on Personal Relationships scale. This validated scale contains 4 items to which responders are asked to indicate their level of agreement over the previous year on a 5-point Likert scale (0=not at all true;4=completely true). The scale score is calculated by determining the mean 0-4 score across the 4 items and normalizing the score to 0-10 scale with higher scores indicating worse outcomes (more adverse impact of work on personal relationships)
Postpartum Depression Screening | At enrollment and at 16 weeks postpartum
  Edinburgh Postnatal Depression Scale. This validated scale includes 10 short statements to which respondents indicate their level of agreement in the past week. Each question is scored from 0-3 and the total score is found by adding the scores from each of the 10 items. The range of the scale is 0-30 with higher scores indicating worse outcome (higher likelihood of postpartum depression)
Ability to Meet Breastfeeding Goals | 24 weeks postpartum
  Participants will be asked to answer the survey question, "Did you feel that you achieved your breastfeeding goal?". Participants will be able to respond "yes", "no", and "I am still breastfeeding and not sure if I will achieve my goal yet". Respondents who reply "no" indicate a worse outcome as they were unable to reach their personal goals for duration of breastfeeding.
Duration of Breastfeeding | 24 weeks postpartum
  measured in months
Serious thoughts of quitting training program | At enrollment, 16 weeks postpartum, and 24 weeks postpartum
  Participants will be asked to indicate their level of agreement (1: strongly agree; 5: strongly disagree) to the following statement: "I have considered leaving my program in the last year (due to the experience of pregnancy/parenthood in my current training specialty". Lower score indicates a worse outcome
Regret for a Medical Career | At enrollment, 16 weeks postpartum and 24 weeks postpartum
  Participants will be asked to indicate their level of agreement (1: strongly agree; 5: strongly disagree) with the following statement: "If I could choose again, I would choose a non-medical career more accommodating of parenthood". Lower score indicates a worse outcome
Regret for a Chosen Specialty | At enrollment, 16 weeks postpartum, and 24 weeks postpartum
  Participants will be asked to indicate their level of agreement (1: strongly agree; 5: strongly disagree) with the following statement: "If I could choose again, I would stay in medicine but choose a specialty more accommodating of parenthood than my current specialty". Lower score indicates a worse outcome
Nightly wakenings | Daily for one week after enrollment, then daily from delivery date until 24 weeks postpartum
  The total number of minutes spent awake per sleep episode will be measured by a wearable Fitbit
Nightly sleep duration | Daily for one week after enrollment, then daily from delivery date until 24 weeks postpartum
  The total number of minutes spent asleep per 24 hours will be measured by a wearable Fitbit
Fatigue | 4 weeks, 12 weeks, 16 weeks, 20 weeks, and 24 weeks postpartum
  Adult 8-item Patient Reported Outcomes Measurement Information System (PROMIS) Sleep -Related Impairment Scale.The sleep-related impairment items assess sleepiness during the day and perceived effects on performance in the past 7 days. The scale items are scored on a 5-point Likert scale indicating intensity from "not at all" to "very much," and the raw scores range from 8 to 40 with high scores indicating worse outcomes (more fatigue).

OTHER OUTCOMES:
Burnout measured by emotional exhaustion and Interpersonal Disengagement components of the Stanford Professional Fulfillment Index | 12 months postpartum
  Burnout measured by emotional exhaustion and depersonalization components of the Emotional exhaustion and Interpersonal Disengagement are EACH scored on a scale of 0-10; The Emotional Exhaustion and Interpersonal Disengagement Scores are then averaged for score 0-10. Higher scores indicate higher likelihood of emotional exhaustion, interpersonal disengagement, and burnout (higher score is worse outcome)
Professional Fulfillment measured by the Stanford Professional Fulfillment Index | 12 months postpartum
  Professional Fulfillment is score on a scale of 0-10 with higher scores indicating a higher likelihood of professional fulfillment (higher score is better outcome)
Organization and personal values alignment | 12 months postpartum
  3-item Stanford Values Alignment Scale. This validated instrument contains 3 statements with which participants are asked to indicate their agreement on a 5-point Likert Scale (0=not at all true; 4=completely true). Aggregate scores are determined by summing the 0-4 score of the individual items to yield a total score ranging from 0-12. Higher values are positive (indicate better alignment between organizational and personal values).
Negative Impact of Work on Personal Relationships | 12 months postpartum
  4-item Impact of Work on Personal Relationships scale. This validated scale contains 4 items to which responders are asked to indicate their level of agreement over the previous year on a 5-point Likert scale (0=not at all true;4=completely true). The scale score is calculated by determining the mean 0-4 score across the 4 items and normalizing the score to 0-10 scale with higher scores indicating worse outcomes (more adverse impact of work on personal relationships)
Ability to meet breastfeeding goals | 12 months postpartum
  Participants will be asked to answer the survey question, "Did you feel that you achieved your breastfeeding goal?". Participants will be able to respond "yes", "no", and "I am still breastfeeding and not sure if I will achieve my goal yet". Respondents who reply "no" indicate a worse outcome as they were unable to reach their personal goals for duration of breastfeeding.
Duration of breastfeeding | 12 months postpartum
  measured in months
Serious thoughts of quitting training program | 12 months postpartum
  articipants will be asked to indicate their level of agreement (1: strongly agree; 5: strongly disagree) to the following statement: "I have considered leaving my program in the last year (due to the experience of pregnancy/parenthood in my current training specialty". Lower score indicates a worse outcome
Regret for a Medical Career | 12 months postpartum
  Participants will be asked to indicate their level of agreement (1: strongly agree; 5: strongly disagree) with the following statement: "If I could choose again, I would choose a non-medical career more accommodating of parenthood". Lower score indicates a worse outcome
Regret for a Chosen Specialty | 12 months postpartum
  Participants will be asked to indicate their level of agreement (1: strongly agree; 5: strongly disagree) with the following statement: "If I could choose again, I would stay in medicine but choose a specialty more accommodating of parenthood than my current specialty". Lower score indicates a worse outcome

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared as this it contains sensitive information that is best presented in aggregate to ensure anonymity of participants

REFERENCES:
- [Background] Rangel EL, Castillo-Angeles M, Easter SR, Atkinson RB, Gosain A, Hu YY, Cooper Z, Dey T, Kim E. Incidence of Infertility and Pregnancy Complications in US Female Surgeons. JAMA Surg. 2021 Oct 1;156(10):905-915. doi: 10.1001/jamasurg.2021.3301. PMID 34319353
- [Background] Rangel EL, Smink DS, Castillo-Angeles M, Kwakye G, Changala M, Haider AH, Doherty GM. Pregnancy and Motherhood During Surgical Training. JAMA Surg. 2018 Jul 1;153(7):644-652. doi: 10.1001/jamasurg.2018.0153. PMID 29562068
- [Background] Rangel EL, Lyu H, Haider AH, Castillo-Angeles M, Doherty GM, Smink DS. Factors Associated With Residency and Career Dissatisfaction in Childbearing Surgical Residents. JAMA Surg. 2018 Nov 1;153(11):1004-1011. doi: 10.1001/jamasurg.2018.2571. PMID 30073246
- [Background] Castillo-Angeles M, Smink DS, Rangel EL. Perspectives of US General Surgery Program Directors on Cultural and Fiscal Barriers to Maternity Leave and Postpartum Support During Surgical Training. JAMA Surg. 2021 Jul 1;156(7):647-653. doi: 10.1001/jamasurg.2021.1807. PMID 34009280
- [Background] West CP, Dyrbye LN, Shanafelt TD. Physician burnout: contributors, consequences and solutions. J Intern Med. 2018 Jun;283(6):516-529. doi: 10.1111/joim.12752. Epub 2018 Mar 24. PMID 29505159
- [Background] Dyrbye LN, West CP, Satele D, Boone S, Tan L, Sloan J, Shanafelt TD. Burnout among U.S. medical students, residents, and early career physicians relative to the general U.S. population. Acad Med. 2014 Mar;89(3):443-51. doi: 10.1097/ACM.0000000000000134. PMID 24448053
- [Background] Dyrbye LN, Freischlag J, Kaups KL, Oreskovich MR, Satele DV, Hanks JB, Sloan JA, Balch CM, Shanafelt TD. Work-home conflicts have a substantial impact on career decisions that affect the adequacy of the surgical workforce. Arch Surg. 2012 Oct;147(10):933-9. doi: 10.1001/archsurg.2012.835. PMID 23117833
- [Background] Stack SW, McKinney CM, Spiekerman C, Best JA. Childbearing and maternity leave in residency: determinants and well-being outcomes. Postgrad Med J. 2018 Dec;94(1118):694-699. doi: 10.1136/postgradmedj-2018-135960. Epub 2018 Dec 15. PMID 30554173
- [Background] Dyrbye LN, Burke SE, Hardeman RR, Herrin J, Wittlin NM, Yeazel M, Dovidio JF, Cunningham B, White RO, Phelan SM, Satele DV, Shanafelt TD, van Ryn M. Association of Clinical Specialty With Symptoms of Burnout and Career Choice Regret Among US Resident Physicians. JAMA. 2018 Sep 18;320(11):1114-1130. doi: 10.1001/jama.2018.12615. PMID 30422299
- [Background] Sandler BJ, Tackett JJ, Longo WE, Yoo PS. Pregnancy and Parenthood among Surgery Residents: Results of the First Nationwide Survey of General Surgery Residency Program Directors. J Am Coll Surg. 2016 Jun;222(6):1090-6. doi: 10.1016/j.jamcollsurg.2015.12.004. Epub 2015 Dec 18. PMID 26776357
- [Background] Melnitchouk N, Scully RE, Davids JS. Barriers to Breastfeeding for US Physicians Who Are Mothers. JAMA Intern Med. 2018 Aug 1;178(8):1130-1132. doi: 10.1001/jamainternmed.2018.0320. PMID 29554184
- [Background] Peters GW, Kuczmarska-Haas A, Holliday EB, Puckett L. Lactation challenges of resident physicians- results of a national survey. BMC Pregnancy Childbirth. 2020 Dec 9;20(1):762. doi: 10.1186/s12884-020-03436-3. PMID 33297993
- [Background] Kancherla BS, Upender R, Collen JF, Rishi MA, Sullivan SS, Ahmed O, Berneking M, Flynn-Evans EE, Peters BR, Gurubhagavatula I. What is the role of sleep in physician burnout? J Clin Sleep Med. 2020 May 15;16(5):807-810. doi: 10.5664/jcsm.8412. Epub 2020 Feb 28. PMID 32108567
- [Background] Ekstedt M, Soderstrom M, Akerstedt T. Sleep physiology in recovery from burnout. Biol Psychol. 2009 Dec;82(3):267-73. doi: 10.1016/j.biopsycho.2009.08.006. Epub 2009 Aug 21. PMID 19699775
- [Background] Lyu HG, Davids JS, Scully RE, Melnitchouk N. Association of Domestic Responsibilities With Career Satisfaction for Physician Mothers in Procedural vs Nonprocedural Fields. JAMA Surg. 2019 Aug 1;154(8):689-695. doi: 10.1001/jamasurg.2019.0529. PMID 30969336
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Livingston-Rosanoff D, Shubeck SP, Kanters AE, Dossett LA, Minter RM, Wilke LG. Got Milk? Design and Implementation of a Lactation Support Program for Surgeons. Ann Surg. 2019 Jul;270(1):31-32. doi: 10.1097/SLA.0000000000003269. No abstract available. PMID 30921050
- [Background] Trockel MT, Menon NK, Rowe SG, Stewart MT, Smith R, Lu M, Kim PK, Quinn MA, Lawrence E, Marchalik D, Farley H, Normand P, Felder M, Dudley JC, Shanafelt TD. Assessment of Physician Sleep and Wellness, Burnout, and Clinically Significant Medical Errors. JAMA Netw Open. 2020 Dec 1;3(12):e2028111. doi: 10.1001/jamanetworkopen.2020.28111. PMID 33284339